CLINICAL TRIAL: NCT02743494
Title: A Randomized, Multicenter, Double Blind, Phase III Study of Adjuvant Nivolumab or Placebo in Subjects With Resected Esophageal, or Gastroesophageal Junction Cancer
Brief Title: An Investigational Immuno-therapy Study of Nivolumab or Placebo in Participants With Resected Esophageal or Gastroesophageal Junction Cancer
Acronym: CheckMate 577
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-577; 2015-005556-10 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Arms: Nivolumab
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether Nivolumab will improve disease-free survival compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Stage II/III carcinoma of the esophagus or gastroesophageal junction
* Completed pre-operative chemo radiotherapy followed by surgery
* Diagnosed with residual pathologic disease after being surgically rendered free of disease with negative margins following complete resection

Exclusion Criteria:

* Diagnosed with cervical esophageal carcinoma
* Diagnosed with Stage IV resectable disease
* Did not receive concurrent chemoradiotherapy prior to surgery
* Participants who have received a live/attenuated vaccine within 30 days of the first treatment

Other protocol defined Inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (204):
- United States (38):
  - Local Institution - 0250, Tucson, Arizona
  - Local Institution - 0026, Los Angeles, California
  - Local Institution - 0023, San Francisco, California
  - Local Institution - 0068, San Francisco, California
  - Local Institution - 0151, Aurora, Colorado
  - Local Institution - 0247, Denver, Colorado
  - Local Institution - 0054, Washington D.C., District of Columbia
  - Local Institution - 0113, Fort Myers, Florida
  - Local Institution - 0131, Jacksonville, Florida
  - Local Institution - 0226, Miami, Florida
  - Local Institution - 0022, Pensacola, Florida
  - Local Institution - 0114, St. Petersburg, Florida
  - Local Institution - 0153, Chicago, Illinois
  - Local Institution - 0025, Baltimore, Maryland
  - Local Institution - 0055, Boston, Massachusetts
  - Local Institution - 0170, Boston, Massachusetts
  - Local Institution - 0171, Boston, Massachusetts
  - Local Institution - 0217, Boston, Massachusetts
  - Local Institution - 0027, St Louis, Missouri
  - Local Institution - 0058, Hackensack, New Jersey
  - Local Institution - 0066, Neptune City, New Jersey
  - Local Institution - 0032, New York, New York
  - Local Institution - 0205, The Bronx, New York
  - Local Institution - 0033, Charlotte, North Carolina
  - Local Institution - 0024, Durham, North Carolina
  - Local Institution - 0056, Cleveland, Ohio
  - Local Institution - 0165, Portland, Oregon
  - Local Institution - 0101, Allentown, Pennsylvania
  - Local Institution - 0048, Philadelphia, Pennsylvania
  - Local Institution - 0116, Pittsburgh, Pennsylvania
  - Local Institution - 0111, Nashville, Tennessee
  - Local Institution - 0130, Nashville, Tennessee
  - Local Institution - 0216, Dallas, Texas
  - Local Institution - 0248, Dallas, Texas
  - Local Institution - 0012, Houston, Texas
  - Local Institution - 0241, Seattle, Washington
  - Local Institution - 0067, Seattle, Washington
  - Local Institution - 0069, Madison, Wisconsin
- Argentina (9):
  - Local Institution - 0050, Capital Federal, Buenos Aires
  - Local Institution - 0152, Capital Federal, Buenos Aires
  - Local Institution - 0164, Ciudad Autonoma Buenos Aires, Distrito Federal
  - Local Institution - 0207, Viedma, Río Negro Province
  - Local Institution - 0208, Rosario, Santa Fe Province
  - Local Institution - 0051, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0198, Buenos Aires
  - Local Institution - 0133, CABA
  - Local Institution - 0112, Córdoba
- Australia (10):
  - Local Institution - 0200, Blacktown, New South Wales
  - Local Institution - 0098, Gosford, New South Wales
  - Local Institution - 0140, Kanwal, New South Wales
  - Local Institution - 0074, St Leonards, New South Wales
  - Local Institution - 0075, Tamworth, New South Wales
  - Local Institution - 0237, Brisbane, Queensland
  - Local Institution - 0123, Adelaide, South Australia
  - Local Institution - 0072, Clayton, Victoria
  - Local Institution - 0156, Perth, Western Australia
  - Local Institution - 0099, Hobart
- Belgium (6):
  - Local Institution - 0035, Brussels
  - Local Institution - 0037, Edegem
  - Local Institution - 0086, Ghent
  - Local Institution - 0034, Leuven
  - Local Institution - 0036, Liège
  - Local Institution - 0087, Namur
- Brazil (12):
  - Local Institution - 0095, Brasília, Federal District
  - Local Institution - 0096, Belo Horizonte, Minas Gerais
  - Local Institution - 0221, Curitiba, Paraná
  - Local Institution - 0059, Ijuí, Rio Grande do Sul
  - Local Institution - 0060, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0223, Itacorubi, Florianopolis, Santa Catarina
  - Local Institution - 0061, Barretos, São Paulo
  - Local Institution - 0222, Sao Jose de Rio Preto, São Paulo
  - Local Institution - 0065, Rio de Janeiro
  - Local Institution - 0064, Salvador
  - Local Institution - 0062, São Paulo
  - Local Institution - 0063, São Paulo
- Canada (9):
  - Local Institution - 0129, Edmonton, Alberta
  - Local Institution - 0093, Vancouver, British Columbia
  - Local Institution - 0092, Halifax, Nova Scotia
  - Local Institution - 0094, London, Ontario
  - Local Institution - 0091, Ottawa, Ontario
  - Local Institution - 0110, Toronto, Ontario
  - Local Institution - 0134, Montreal, Quebec
  - Local Institution - 0109, Québec, Quebec
  - Local Institution - 0214, Trois-Rivières, Quebec
- China (9):
  - Local Institution - 0240, Beijing, Beijing Municipality
  - Local Institution - 0234, Fuzhou, Fujian
  - Local Institution - 0227, Shanghai, Shanghai Municipality
  - Local Institution - 0239, Shanghai, Shanghai Municipality
  - Local Institution - 0230, Hangzhou, Zhejiang
  - Local Institution - 0238, Hangzhou, Zhejiang
  - Local Institution - 0233, Linhai, Zhejiang
  - Local Institution - 0232, Shanghai
  - Local Institution - 0228, Tianjin
- Czechia (3):
  - Local Institution - 0031, Brno
  - Local Institution - 0029, Hradec Králové
  - Local Institution - 0030, Olomouc
- Local Institution - 0166, Aarhus N, Central Jutland, Denmark
- France (9):
  - Local Institution - 0215, Avignon Cedes 9
  - Local Institution - 0121, Dijon
  - Local Institution - 0117, Lille
  - Local Institution - 0119, Paris
  - Local Institution - 0120, Pessac
  - Local Institution - 0118, Pierre-Bénite
  - Local Institution - 0132, Rennes
  - Local Institution - 0149, Rouen
  - Local Institution - 0148, Toulouse
- Germany (8):
  - Local Institution - 0001, Mainz, Rhineland-Palatinate
  - Local Institution - 0006, Berlin
  - Local Institution - 0003, Cologne
  - Local Institution - 0008, Essen
  - Local Institution - 0007, Hamburg
  - Local Institution - 0017, Marburg
  - Local Institution - 0005, Munich
  - Local Institution - 0011, Tübingen
- Local Institution - 0225, Hong Kong, Hong Kong
- Hungary (4):
  - Local Institution - 0053, Budapest
  - Local Institution - 0224, Budapest
  - Local Institution - 0052, Debrecen
  - Local Institution - 0057, Kaposvár
- Ireland (3):
  - Local Institution - 0039, Wilton, CORK
  - Local Institution - 0040, Dublin
  - Local Institution - 0038, Galway
- Israel (5):
  - Local Institution - 0146, Haifa
  - Local Institution - 0144, Jerusalem
  - Local Institution - 0143, Petah Tikva
  - Local Institution - 0145, Ramat Gan
  - Local Institution - 0142, Tel Aviv
- Italy (5):
  - Local Institution - 0105, Bergamo
  - Local Institution - 0137, Milan
  - Local Institution - 0104, Milan
  - Local Institution - 0106, Reggio Emilia
  - Local Institution - 0107, Roma
- Japan (20):
  - Local Institution - 0173, Akita, Akita
  - Local Institution - 0180, Chiba, Chiba
  - Local Institution - 0187, Fukuoka, Fukuoka
  - Local Institution - 0189, Gifu, Gifu
  - Local Institution - 0183, Hiroshima, Hiroshima
  - Local Institution - 0192, Sapporo, Hokkaido
  - Local Institution - 0196, Sapporo, Hokkaido
  - Local Institution - 0191, Kagoshima, Kagoshima-ken
  - Local Institution - 0184, Kumamoto, Kumamoto
  - Local Institution - 0188, Sendai, Miyagi
  - Local Institution - 0182, Sayama, Osaka
  - Local Institution - 0185, Suita-shi, Osaka
  - Local Institution - 0186, Kitaadachi-gun, Saitama
  - Local Institution - 0172, Chuo-ku, Tokyo
  - Local Institution - 0190, Koto-ku, Tokyo
  - Local Institution - 0174, Minato-ku, Tokyo
  - Local Institution - 0193, Shinjuku-ku, Tokyo
  - Local Institution - 0204, Shinjuuku-ku, Tokyo
  - Local Institution - 0194, Fukuoka
  - Local Institution - 0181, Kita-gun
- Mexico (6):
  - Local Institution - 0212, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 0085, Tlalpan, Distrito Federal C.p.
  - Local Institution - 0127, Leon, Guanajato, Guanajuato
  - Local Institution - 0154, Aguascalientes
  - Local Institution - 0084, Distrito Federal
  - Local Institution - 0168, Mexico City
- Netherlands (3):
  - Local Institution - 0089, Amsterdam, North Holland
  - Local Institution - 0042, Groningen
  - Local Institution - 0043, Maastrict
- Peru (4):
  - Local Institution - 0195, Callao
  - Local Institution - 0162, Lima
  - Local Institution - 0141, Lima
  - Local Institution - 0088, Lima
- Poland (5):
  - Local Institution - 0083, Gliwice
  - Local Institution - 0138, Krakow
  - Local Institution - 0139, Lublin
  - Local Institution - 0082, Poznan
  - Local Institution - 0081, Warsaw
- Local Institution - 0097, San Juan, Puerto Rico
- Romania (6):
  - Local Institution - 0167, Baia Mare
  - Local Institution - 0197, Bucharest
  - Local Institution - 0163, Bucharest
  - Local Institution - 0103, Cluj-Napoca
  - Local Institution - 0028, Craiova
  - Local Institution - 0135, Floreşti
- Russia (4):
  - Local Institution - 0213, Cheboksary
  - Local Institution - 0125, Moscow
  - Local Institution - 0209, Saint Petersburg
  - Local Institution - 0136, Saint Petersburg
- Singapore (2):
  - Local Institution - 0219, Singapore, Central Singapore
  - Local Institution - 0218, Singapore
- South Korea (2):
  - Local Institution - 0175, Songpa-gu, Seoul
  - Local Institution - 0176, Seoul
- Spain (4):
  - Local Institution - 0078, Barcelona
  - Local Institution - 0079, Córdoba
  - Local Institution - 0080, Madrid
  - Local Institution - 0077, Madrid
- Switzerland (2):
  - Local Institution - 0018, Basel
  - Local Institution - 0047, Sankt Gallen
- Taiwan (3):
  - Local Institution - 0177, Taichung
  - Local Institution - 0178, Tainan
  - Local Institution - 0179, Taipei
- Turkey (Türkiye) (3):
  - Local Institution - 0160, Adana
  - Local Institution - 0161, Erzurum
  - Local Institution - 0157, Istanbul
- United Kingdom (7):
  - Local Institution - 0203, London, Greater London
  - Local Institution - 0045, London, Greater London
  - Local Institution - 0046, Southampton, Hampshire
  - Local Institution - 0049, Withington, Manchester
  - Local Institution - 0169, Sutton, Surrey
  - Local Institution - 0243, Cardiff
  - Local Institution - 0202, London

REFERENCES:
- [Derived] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 794 participants were randomized and 792 were treated. The reasons for the 2 participants not being treated were: Participant request to discontinue study treatment (1) and Participant no longer meeting study criteria (1).
Groups:
- Nivolumab: Nivolumab 240 mg Q2W for 8 cycles (16 weeks) followed by Nivolumab 480 mg Q4W for 9 cycles.
- Placebo: Placebo IV Q2W for 8 cycles (16 weeks) followed by Placebo IV Q4W for 9 cycles
Period: Pre-treatment Period
Arm/Group | Nivolumab | Placebo
Started (Started = randomized) | 532 | 262
Completed (Completed = Entering the treatment period) | 532 | 260
Not Completed | 0 | 2
Not completed — Participant request to discontinue treatment | 0 | 1
Not completed — Participant no longer meeting study criteria | 0 | 1
Period: Treatment Period
Arm/Group | Nivolumab | Placebo
Started | 532 | 260
Completed | 260 | 116
Not Completed | 272 | 144
Not completed — Disease recurrence | 152 | 115
Not completed — Study drug toxicity | 56 | 8
Not completed — Death | 1 | 1
Not completed — Adverse event unrelated to study drug | 15 | 9
Not completed — Participant request to discontinue treatment | 31 | 5
Not completed — Participant withdrew consent | 11 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Poor/Non-compliance | 2 | 0
Not completed — Other reasons | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Placebo | Total
Number analyzed (Participants) | 532 | 262 | 794
Age, Continuous [Mean (Standard Deviation); unit: Years] — All randomized participants
  Years | 60.8 (9.2) | 59.9 (10.1) | 60.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — All randomized participants
  Participants
    Female | 83 | 40 | 123
    Male | 449 | 222 | 671
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All randomized participants
  Participants
    Hispanic or Latino | 33 | 11 | 44
    Not Hispanic or Latino | 268 | 144 | 412
    Unknown or Not Reported | 231 | 107 | 338
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 432 | 216 | 648
  Black or African American | 7 | 2 | 9
  Asian | 83 | 34 | 117
  American Indian or Alaska Native | 0 | 2 | 2
  Other | 10 | 7 | 17
  Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival is defined as the time between randomization date and first date of recurrence or death, whichever occurs first.
  Recurrence is defined as the appearance of one or more new lesions, which can be local, regional, or distant in location from the primary resected site ( assessed by imaging or pathology). All deaths without prior recurrence are considered as DFS events. For participants who remained alive and without recurrence, DFS was censured on the date of last evaluable disease assessment
Time Frame: From randomization to the date of recurrence or death (up to approximately 46 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 532 | 262
Months | 22.41 [16.62 to 34.00] | 11.04 [8.34 to 14.32]
Statistical Analysis 1: Comparison: Nivolumab vs Placebo; Test type: Superiority; p = 0.0003, Stratified log-rank test; Hazard Ratio (HR) = 0.69, 96.4% CI 2-sided [0.56 to 0.86] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab over Placebo

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death from any cause. For subjects that are alive, their survival time was censored at the date of last contact date (or "last known alive date"). Overall survival was censored at the date of randomization for subjects who were randomized but had no follow-up.
Time Frame: From randomization to the date of death (up to approximately 60 months)
Population: All randomized participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 532 | 262
Months | 51.71 [41.03 to 61.63] | 35.25 [30.72 to 48.76]
Statistical Analysis 1: Comparison: Nivolumab vs Placebo; Test type: Superiority; p = 0.1064, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.070 to 1.03] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab over Placebo

3. Secondary Outcome: Overall Survival Rates at 12-, 24-, and 36-months
Description: Overall survival rate is defined as the percentage of participants who are alive at 1, 2 and 3 years following randomization
Time Frame: At 12-, 24- and 36-months post first dose.
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 532 | 262
Percent of participants
  12-months | 87.5 [84.4 to 90.0] | 84.6 [79.6 to 88.4]
  24-months | 68.1 [63.9 to 71.9] | 65.8 [59.6 to 71.2]
  36-months | 56.9 [52.5 to 61.0] | 49.7 [43.5 to 55.7]

ADVERSE EVENTS:
Time Frame: All-cause Mortality was collected from randomization until the data cutoff date (up to approximately 60 months). SAEs and Other AEs were collected from the first dose to 30 days following the last dose (an average of 9 months up to a maximum of 16 months).
Description: All-cause mortality represents all randomized participants. Serious adverse events (SAEs) and other adverse events (AEs) represents participants who received at least one dose of study medicine.
Arm/Group | Nivolumab | Placebo
All-Cause Mortality (participants affected / at risk) | 299/532 | 162/262
Serious Adverse Events (participants affected / at risk) | 196/532 | 99/260
Other Adverse Events (participants affected / at risk) | 470/532 | 216/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=532) | Placebo (N=260)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocarditis (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 6
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Fibrosing colonopathy (Gastrointestinal disorders) | 1 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 5 | 2
Ileus (Gastrointestinal disorders) | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 4 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pylorospasm (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Complication associated with device (General disorders) | 0 | 1
Disease recurrence (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Polyserositis (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Sudden death (General disorders) | 2 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Parapharyngeal space infection (Infections and infestations) | 0 | 1
Periumbilical abscess (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 20 | 6
Pneumonia aspiration (Infections and infestations) | 8 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 0 | 1
Subacute endocarditis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 1 | 0
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Product dispensing error (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 | 31
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 2
Facial nerve disorder (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lhermitte's sign (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Device occlusion (Product Issues) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=532) | Placebo (N=260)
Anaemia (Blood and lymphatic system disorders) | 50 | 22
Hyperthyroidism (Endocrine disorders) | 44 | 2
Hypothyroidism (Endocrine disorders) | 67 | 7
Abdominal pain (Gastrointestinal disorders) | 71 | 39
Abdominal pain upper (Gastrointestinal disorders) | 21 | 19
Constipation (Gastrointestinal disorders) | 65 | 36
Diarrhoea (Gastrointestinal disorders) | 165 | 84
Dry mouth (Gastrointestinal disorders) | 28 | 10
Dysphagia (Gastrointestinal disorders) | 68 | 42
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 48 | 36
Nausea (Gastrointestinal disorders) | 129 | 62
Vomiting (Gastrointestinal disorders) | 86 | 42
Asthenia (General disorders) | 43 | 16
Fatigue (General disorders) | 153 | 67
Influenza like illness (General disorders) | 27 | 8
Pyrexia (General disorders) | 34 | 11
Nasopharyngitis (Infections and infestations) | 16 | 14
Pneumonia (Infections and infestations) | 30 | 11
Upper respiratory tract infection (Infections and infestations) | 20 | 15
Alanine aminotransferase increased (Investigations) | 43 | 6
Amylase increased (Investigations) | 28 | 5
Aspartate aminotransferase increased (Investigations) | 51 | 14
Blood alkaline phosphatase increased (Investigations) | 33 | 6
Weight decreased (Investigations) | 75 | 26
Decreased appetite (Metabolism and nutrition disorders) | 87 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 12
Dizziness (Nervous system disorders) | 53 | 24
Headache (Nervous system disorders) | 43 | 30
Insomnia (Psychiatric disorders) | 29 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 106 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 71 | 16
Rash (Skin and subcutaneous tissue disorders) | 66 | 17
Hypertension (Vascular disorders) | 38 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT02743494/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT02743494/SAP_001.pdf